CLINICAL TRIAL: NCT05816824
Title: The Effect of Visual Feedback Based Clinical Monitoring Software on Clinical and Psychosocial Symptoms in Patients With Chronic Low Back Pain
Brief Title: The Effect of Clinical Monitoring Software on Symptoms in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatih Ozden, Assistant Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fizyoanalist
Record Dates: First submitted 2023-03-22; First posted 2023-04-18 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symptom Monitoring Telerehabilitation (Intervention) Group (Experimental): The intervention group will be followed up with the same protocol plus symptom monitoring software called PhysioAnalyst which provides visual feedback. The video exercises given to the participants will include Williams, McKenzie exercises and core strengthening exercises.
  Interventions: Other: Symptom monitoring software via visual feedback
- Telerehabilitation (Control) Group (Active Comparator): The control group will receive video exercise-based rehabilitation protocol with telerehabilitation without visual feedback. The video exercises given to the participants will include Williams, McKenzie exercises and core strengthening exercises.
  Interventions: Other: Symptom monitoring software via visual feedback

INTERVENTIONS:
Other: Symptom monitoring software via visual feedback — With PhysioAnalyst software, individuals are evaluated using clinical tools (questionnaire, scale). These evaluations provide visual feedback to individuals in the form of tables and graphs. In this way, patients can observe the changes in their clinical status.

SUMMARY:
The aim of this randomised controlled trial is to compare the effectiveness of two different telerehabilitation assessment methods in patients with chronic low back pain. The control group will receive a video exercise-based rehabilitation protocol with telerehabilitation. The intervention group will be followed up with the same protocol plus symptom monitoring software called PhysioAnalyst which provides visual feedback. The evaluation of outcome measures will be performed on the control group through the PhysioAnalist programme without visual feedback and on the intervention group through the PhysioAnalist programme with visual feedback.

DETAILED DESCRIPTION:
Individuals with chronic low back pain will be divided into 2 groups by randomisation software (https://ctrandomization.cancer.gov/tool/). The control group will be given video exercises on the online platform. Initial, interim and final evaluations will be performed by filling in the patient-reported outcome measures through the PhysioAnalyst programme without patient feedback. The intervention group will be given the video exercise programme on the same online platform. Initial, intermediate and final assessments will be performed with our self-developed PhysioAnalyst software using visual feedback tools. The video exercises given to the participants will include Williams, McKenzie exercises and core strengthening exercises. Visual Analogue Scale pain score, Nottingham Health Profile, Pain Catastrophising Scale, Oswestry Disability Index, Telehealth Usability Questionnaire, Telemedicine Satisfaction Questionnaire, Exercise Adherence Rating Scale will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with low back pain for more than 3 months and diagnosed with chronic low back pain
* Adult patients aged between 18 and 65 years
* Individuals without a radicular symptom
* Patients who can understand and respond to verbal commands and who do not have hearing or speech problems or psychiatric problems that may prevent communication
* Patients who have devices with sufficient requirements to receive the exercise programme and assessments offered by telerehabilitation

Exclusion Criteria:

* Spinal surgery history
* Presence of malignancy
* Presence of other orthopaedic and/or neurological diseases that may affect the assessment and treatment
* Pregnant women or women with suspected pregnancy
* Patients who did not sign the consent form required for participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-04-30 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-08-05 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Change from Baseline Visual Analog Scale at 8 weeks
  On a 10 cm straight line or numerical and visual scale, the patient is asked to mark the pain felt (0: no pain, 10: unbearable pain).
Nottingham Health Profile | Change from Baseline Nottingham Health Profile at 8 weeks
  The measure consists of six different subcategories testing physical activity, energy, pain, social isolation, sleep and emotional responses. Scores range from 0 to 100 for each subcategory. Low scores indicate a low impact of the complaint and high scores indicate a high impact of the complaint.
Pain Catastrophising Scale | Change from Baseline Pain Catastrophising Scale at 8 weeks
  Scale is used to assess the patient's feelings and thoughts about pain and disaster. The total score ranges from 0 to 52 points. A high score indicates a bad situation.
Oswestry Disability Index | Change from Baseline Oswestry Disability Index at 8 weeks
  The Oswestry Disability Index consists of 10 questions measuring functional status. Each question is evaluated between 0 and 5 points and the total maximum score is 50. Higher score indicates more disability.

SECONDARY OUTCOMES:
Telehealth Usability Questionnaire | Change from Baseline Telehealth Usability Questionnaire at 8 weeks
  The survey addresses six factors; usability, ease of use and learnability, interface quality, interaction quality, reliability and satisfaction. Total score is ranged between 21 to 147. A higher score indicates better usability.
Telemedicine Satisfaction Questionnaire | Change from Baseline Telemedicine Satisfaction Questionnaire at 8 weeks
  Treatment of patients or other remote level of satisfaction with the software or system from which they receive rehabilitation services is being evaluated. The total score ranges between 14-70. A higher score indicates better satisfaction.
Exercise Adherence Rating Scale | Change from Exercise Adherence Rating Scale at 8 weeks
  Exercise Adherence Rating Scale is a self-report measure that is composed of six items that directly assess adherence behavior. Higher scores indicating greater adherence (0 to 24).

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Özden, PhD, Principal Investigator — Muğla Sıtkı Koçman University; Bekir Güçlü, MSc, Study Chair — Istanbul Halic University; İsmet Tümtürk, MSc, Study Chair — Süleyman Demirel University; Ahmet İmerci, MD, Study Chair — Muğla Sıtkı Koçman University; Baki Umut Tuğay, PhD, Study Chair — Muğla Sıtkı Koçman University
Locations (1):
- Muğla Sıtkı Koçman Training and Research Hospital, Muğla, Menteşe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No